CLINICAL TRIAL: NCT03022799
Title: A First in Human, Randomized, Double-blind, Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Following Single and Multiple Oral Doses of KM-819 in Healthy Young Adult and Elderly Subjects
Brief Title: Phase I, KM-819 in Healthy Subjects for Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kainos Medicine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KMCP-819-K101
Record Dates: First submitted 2016-12-27; First posted 2017-01-18 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-03

CONDITIONS: Parkinson's Disease
Keywords: FAF1; Fas (TNFRSF6)-associated factor 1; FAF1 inhibitor; KM-819
MeSH Terms: conditions — Parkinson Disease; Autoimmune Lymphoproliferative Syndrome, Type IA | interventions — KM-819

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KM-819 (Experimental): Each cohort consists of 8 subjects; 6 subjects will receive planned dose of KM-819 and 2 subjects will receive placebo.
  Interventions: Drug: KM-819
- Placebo (Placebo Comparator): Each cohort consists of 8 subjects; 6 subjects will receive planned dose of KM-819 and 2 subjects will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KM-819
  Arms: KM-819
Drug: Placebo
  Arms: Placebo

SUMMARY:
This first in human, single-center, randomized, placebo-controlled, double blind, sequential group Phase 1 study in healthy subjects will be conducted to evaluate the safety, tolerability, PK, and PD following the escalation of single and multiple doses of KM-819.

The study will consist of 2 parts. In Part A, up to 5 cohorts of young adult male subjects, and 1 single dose cohort of elderly male or post menopausal female subjects will receive escalating single doses of KM-819. In Part B, up to 4 cohorts of healthy young adult male subjects and 1 multiple dose cohort of elderly male or post menopausal female subjects will receive escalating multiple doses of KM-819. Part B will be conducted after completion of all cohorts of young adult male subjects in Part A.

Dose escalation to the next level will be determined using safety, tolerability, and PK data of the previous cohort.

Part A, Single Ascending Dose (SAD) Up to 40 healthy young adult male subjects and 8 healthy elderly male or post menopausal female subjects will be enrolled and randomized to receive either KM-819 or placebo.

Each of the 5 dose escalation cohorts consists of 8 healthy young adult male subjects; 6 subjects will receive 10, 30, 100, 200, or 400 mg of KM-819 and 2 subjects will receive placebo. In each single dose cohort, dosing of subjects will be sentinel, i.e., 2 subjects will be dosed on the first day (1 subject will receive active treatment and 1 subject will receive placebo) and the remaining 6 subjects will be dosed at least 24 hours after the first 2 subjects.

Cohorts will be dosed sequentially with escalating doses. Eight elderly male or post-menopausal female subjects will be enrolled into an additional cohort; 6 subjects will receive 200 mg KM-819 and 2 subjects will receive placebo.

Part A consists of a Screening period of up to 28 days, and a 3 day Confinement period when subjects are hospitalized for study activities. Subjects are required to return for outpatient visits on Day 4, 7 and for the Follow up Visit on Day 14.

Part B, Multiple Ascending Dose (MAD) Up to 32 healthy young adult male subjects and 8 healthy elderly male or post menopausal female subjects will be enrolled and randomized to receive either KM-819 or placebo.

Each of the 4 dose escalation cohorts consists of 8 healthy young adult male subjects; 6 subjects will receive 30, 100, 200, or 400 mg of KM-819 once a day (QD) for 7 days and 2 subjects will receive placebo. Cohorts will be dosed sequentially with escalating doses.

Eight elderly male or post-menopausal female subjects will be enrolled into an additional cohort; 6 subjects will receive 200 mg KM-819 QD for 7 days and 2 subjects will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written informed consent and privacy language as per national regulations must be obtained from the subject prior to any study-related procedures (including withdrawal of prohibited medication, if applicable).
2. Male subject should be 19 to 45 years old (for young adult cohorts) or over 60 years old (for elderly cohorts).
3. Subject has a body mass index (BMI) range of 18.5 to 30 kg/m2 inclusive at Screening.
4. Male subject and his female spouse/partner who is of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (at least one of which must be a barrier method) starting at Screening and continuing throughout the study period and for 90 days after final study drug administration. Highly effective contraception is defined as:

   * Established use of oral, injected, or implanted hormonal methods of contraception
   * Placement of an intrauterine device or intrauterine system
   * Barrier methods of contraception: condom with spermicidal foam, gel, film, cream, suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam, gel, film, cream, or suppository
5. Male subject must not donate sperm starting at Screening, throughout the study period and for at least 90 days after final study drug administration.
6. Female subject must be over 60 years old and post-menopausal (defined as at least 1 year without any menses) prior to Screening.
7. Subject agrees not to participate in another investigational study while on study treatment.

Exclusion Criteria:

1. Subject has a known or suspected hypersensitivity to KM-819, or any components of the formulation(s) used.
2. Subject has previously participated in a clinical study with KM-819.
3. Subject has any of the liver enzymes (aspartate aminotransferase [AST], alanine transaminase [ALT], alkaline phosphatase, γ glutamyl transferase) or total bilirubin (TBIL) above the ULN. If any liver enzyme is > 1 × ULN but < 1.5 × ULN, the assessment may be repeated once during the Screening period or on check-in. If the repeated assessment is above the ULN, it is exclusionary. If the initial value is > 1.5 × ULN, it cannot be repeated and is exclusionary.
4. Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, allergic rhinitis or rhino-conjunctivitis, or house dust mite allergy at time of dosing).
5. Subject with a history of a suicide attempt or suicidal behavior. Any recent suicidal ideation (a level of 4 or 5) within the last 3 months, or having a positive C-SSRS at check-in (Day -1), or who is at significant risk to commit suicide, as judged by the Investigator using the C SSRS at Screening.
6. Subject has/had febrile illness or symptomatic viral, bacterial (including upper respiratory infection) or fungal (non-cutaneous) infection within 1 week before site check-in.
7. Subject has any clinically significant abnormality following the Investigator's review of the physical examination, ECG, and protocol-defined clinical laboratory tests at Screening or site check-in.
8. Subject has a mean pulse < 40 or > 90 beats per minute (bpm); mean systolic blood pressure (SBP) > 140 mmHg; or mean diastolic blood pressure (DBP) > 90 mmHg (measurements taken in triplicate after subject has been resting in the supine position for 5 minutes; pulse will be measured automatically) at Screening or check-in. If the mean pulse, mean SBP, or mean DBP is out of the range specified above, 1 additional triplicate measurement may be taken at Screening and check-in.
9. Subject has a mean QTcF interval of > 430 msec (for males) and > 450 msec (for females) at Screening or check-in. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken. If this triplicate also gives an abnormal result, the subject should be excluded.
10. Subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsade de pointes, structural heart disease, or a family history of Long QT Syndrome.
11. Subject has use of any prescribed or non-prescribed drugs (including vitamins, hormone replacement therapy, natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks before study drug administration. Acetaminophen up to 2000 mg/day is allowed.
12. Subject has had any use of tobacco- or nicotine-containing products within 6 months prior to Screening.
13. Subject has history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to Screening or has a history of alcoholism or abuse of amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates (drugs-of-abuse) within the past 2 years prior to Screening (Note: 1 unit = 355 mL of beer, 118 mL of wine, or 29 mL of spirits/hard liquor) or the subject tests positive at Screening or site admission for alcohol or drugs of-abuse.
14. Subject has used any drugs-of-abuse within 3 months before check in.
15. Subject has used any inducers of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to check-in.
16. Subject has any significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood, or blood products within 60 days or donated plasma within 7 days before check-in.
17. Subject has a positive serology test for hepatitis B surface antigen (HbsAg), anti hepatitis A virus Immunoglobulin M (HAV IgM), anti-hepatitis C virus (HCV Ab), or anti-human immunodeficiency virus (HIV Ab).
18. Subject has participated in any interventional clinical study or has been treated with any investigational drugs within 3 months or 5 half lives, whichever is longer, before the initiation of Screening.
19. Subject has (recent history of) any other condition which, in the opinion of the Investigator, precludes the subject's participation in the trial.
20. Subject is an employee of the Kainos Medicine, Inc. or vendors involved in the study.

    Additional Exclusion Criteria for Young Adult Subjects
21. For young adult cohorts, subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy, as judged by the Investigator or designee.

Exclusion Criteria for Elderly Subjects Replacement for Exclusion No. 8 above 8. Subject has a mean pulse < 50 or > 90 bpm; mean SBP > 160 mmHg; mean DBP > 100 mmHg (measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically).

Replacement for Exclusion No. 21 above 21. For elderly cohorts, subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy that is not well managed and stable, as judged by the Investigator or designee.

Additional Exclusion Criteria 22. Elderly subject is excluded if the Glomerular Filtration Rate (calculated based on Cockcroft-Gault formula) is < 60 mL/min/1.73 m2.

23. Clinically significant abnormal findings in the lumbar X-ray examination (only for elder subjects for MAD study).

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Moon Lee, PhD, Study Director — Kainos Medicine Inc.
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Individual identifiable personal information will not be shared. All individuals will be coded by a 4-digit study code.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A first in human, single center, randomized, placebo controlled, double blind, sequential group Phase 1 study in healthy subjects recruited from Nov 2016 to Sep 2017. Participants who met all the inclusion and none of the exclusion criteria were enrolled.
Pre-assignment Details: All subjects underwent a Screening period of up to 28 days and a 3 day Confinement period when they were hospitalized for study activities (Day -1 to Day 3) for Part A (Single Ascending Doses) and an 8 day Confinement period when they were hospitalized for study activities (Day -1 to Day 8) for Part B (Multiple Ascending Doses)
Groups:
- KM-819 - 10 mg (Part A): 6 subjects in this cohort received 10 mg of KM-819 orally with approximately 240 mL of water (room temperature), after an overnight fasting for a minimum of 8 hours.
- KM-819 - 30 mg (Part A): 6 subjects in this cohort received 30 mg of KM-819 orally with approximately 240 mL of water (room temperature), after an overnight fasting for a minimum of 8 hours.
- KM-819 - 100mg (Part A): 6 subjects in this cohort received 100 mg of KM-819 orally with approximately 240 mL of water (room temperature), after an overnight fasting for a minimum of 8 hours.
- KM-819 200mg (Part A): 6 subjects in this cohort received 200 mg of KM-819 orally with approximately 240 mL of water (room temperature), after an overnight fasting for a minimum of 8 hours.
- KM-819 - 400mg (Part A): 6 subjects in this cohort received 400 mg of KM-819 orally with approximately 240 mL of water (room temperature), after an overnight fasting for a minimum of 8 hours.
- KM-819 200mg (Elderly Male Subjects) (Part A): 6 elderly male subjects in this cohort received 200 mg of KM-819 orally with approximately 240 mL of water (room temperature), after an overnight fasting for a minimum of 8 hours.
- Placebo (Part A): 12 subjects received placebo orally with approximately 240 mL of water (room temperature), after an overnight fasting for a minimum of 8 hours.
- KM-819 30 mg (Part B): 6 subjects in this cohort received 30 mg of KM-819 orally on Day 2 to Day 6, the study drug was administered with approximately 240 mL of water (room temperature), after an overnight fasting for a minimum of 8 hours.
- KM-819 100 mg (Part B): 6 subjects in this cohort received 100 mg of KM-819 orally on Day 2 to Day 6, the study drug was administered with approximately 240 mL of water (room temperature), after an overnight fasting for a minimum of 8 hours.
- KM-819 200mg (Part B): 6 subjects in this cohort received 200 mg of KM-819 orally on Day 2 to Day 6, the study drug was administered with approximately 240 mL of water (room temperature), after an overnight fasting for a minimum of 8 hours.
- KM-819 400mg (Part B): 6 subjects in this cohort received 400 mg of KM-819 orally on Day 2 to Day 6, the study drug was administered with approximately 240 mL of water (room temperature), after an overnight fasting for a minimum of 8 hours.
- KM-819 200mg (Elderly Male Subjects) (Part B): 6 elderly male subjects in this cohort received 30 mg of KM-819 orally on Day 2 to Day 6, the study drug was administered with approximately 240 mL of water (room temperature), after an overnight fasting for a minimum of 8 hours.
- Placebo (Part B): 10 subjects received placebo of KM-819 orally on Day 2 to Day 6, the study drug was administered with approximately 240 mL of water (room temperature), after an overnight fasting for a minimum of 8 hours.
Period: Overall Study
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | Placebo (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B) | Placebo (Part B)
Started | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 10
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 5 | 5 | 6 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | Placebo (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B) | Placebo (Part B) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 10 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.7 (6.28) | 25.2 (7.57) | 26.2 (5.04) | 27.5 (6.38) | 26.3 (4.13) | 75.0 (5.76) | 35.6 (19.76) | 27.5 (7.56) | 30.2 (6.85) | 28.7 (5.65) | 22.5 (1.38) | 72.8 (6.59) | 38.5 (19.73) | 35.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 10 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 6 | 6 | 6 | 6 | 6 | 6 | 11 | 6 | 6 | 6 | 6 | 6 | 10 | 87
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: All AEs will be coded using the latest available version 19.1 of the Medical Dictionary for Regulatory Activities (MedDRA).
  A treatment-emergent adverse event (TEAE) is defined as an AE that begins or that worsens in severity after at least one dose of the study drug has been administered.
Time Frame: From screening (Day-28 to Day -2), Day -1 to Day 4, Day 7, and follow-up visit Day 14.
Population: All subjects who received at least one dose.
Measure: Number; unit: participants
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | Placebo (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B) | Placebo (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 10
participants
  TEAEs | 2 | 2 | 2 | 1 | 0 | 2 | 3 | 2 | 4 | 5 | 5 | 3 | 5
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Severe TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Related TEAEs | 2 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 2 | 5 | 4 | 3 | 5
  TEAEs leading to withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  TEAEs leading to death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Cmax (Maximum Plasma Concentration Determined Directly From the Concentration-time Profile)
Description: To evaluate Cmax of single and multiple ascending oral doses of KM-819 in healthy young adult male subjects and multiple oral doses of KM-819 in elderly male subjects.
Time Frame: Part A: Day1 to Day 4. Part B: Day-1 to Day 8
Population: All subjects who received at least one dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 244.1 (31.4) | 503.6 (28.0) | 1152 (36.7) | 1879 (55.3) | 2767 (43.4) | 1766 (26.0) | 512.0 (30.9) | 1009 (33.0) | 1465 (77.2) | 3163 (50.7) | 3542 (76.4)

3. Secondary Outcome: Tmax (Time to Achieve Maximum Observed Plasma Concentration Determined Directly From the Concentration-time Profile)
Description: To evaluate the pharmacokinetics and pharmacodynamics of single and multiple ascending oral doses of KM-819 in healthy young adult male subjects and multiple oral doses of KM-819 in elderly male subjects.
Time Frame: Part A:Day 1 to 4; Part B: Day 1 to Day 8
Population: All subjects who received at least one dose.
Measure: Median (Full Range); unit: hours
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours
  Part A: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
  Part A | 1.500 [0.50 to 2.00] | 1.000 [0.50 to 2.00] | 2.000 [1.00 to 4.00] | 2.008 [1.00 to 4.00] | 4.000 [2.00 to 4.00] | 2.000 [1.00 to 4.00] |  |  |  |  |
  Part B-Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Part B-Day 1 |  |  |  |  |  |  | 2.000 [1.00 to 6.00] | 2.000 [1.00 to 4.00] | 3.000 [2.00 to 6.00] | 2.008 [1.00 to 6.00] | 2.000 [1.00 to 6.00]
  Part B-Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Part B-Day 7 |  |  |  |  |  |  | 2.000 [0.97 to 6.00] | 3.000 [1.00 to 4.00] | 4.000 [3.92 to 4.03] | 2.000 [0.50 to 4.00] | 2.017 [1.00 to 4.02]

4. Secondary Outcome: t½ (Apparent Terminal Elimination Half Life)
Description: To evaluate the pharmacokinetics and pharmacodynamics of single and multiple ascending oral doses of KM-819 in healthy young adult male subjects. To evaluate the PK and PD of single and multiple oral doses of KM-819 in elderly male subjects.
Time Frame: Part A: Day 1 to Day 4. Part B: Day1 to Day 8
Population: All subjects who received at least one dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours
  Part A: number analyzed (Participants) | 6 | 6 | 4 | 5 | 5 | 6 | 0 | 0 | 0 | 0 | 0
  Part A | 1.786 (28.3) | 4.791 (25.0) | 9.159 (41.2) | 9.010 (71.6) | 8.527 (63.2) | 10.55 (28.5) |  |  |  |  |
  Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0 | 6
  Part B |  |  |  |  |  |  | 3.075 (46.9) | 5.417 (15.1) | 5.785 (24.1) |  | 4.389 (13.4)

5. Secondary Outcome: Tlag (Lag Time)
Description: To evaluate the T lag of single and multiple ascending oral doses of KM-819 in healthy young adult male subjects and multiple oral doses of KM-819 in elderly male subjects.
Time Frame: Part A: Day1 to Day 4. Part B: Day 1 to Day 8
Population: All subjects who received at least one dose.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours
  Part A: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
  Part A | 0.08333 (0.1291) | 0 (0) | 0 (0) | 0.04167 (0.1021) | 0 (0) | 0 (0) |  |  |  |  |
  Part B-Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Part B-Day 1 |  |  |  |  |  |  | 0.04167 (0.1021) | 0.08333 (0.1291) | 0 (0) | 0 (0) | 0 (0)
  Part B-Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 5 | 5 | 6
  Part B-Day 7 |  |  |  |  |  |  | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

6. Secondary Outcome: AUClast (Area Under the Plasma Concentration-time From Predose (Time 0) to the Last Quantifiable Concentration)
Description: To evaluate AUClast of single and multiple ascending oral doses of KM-819 in healthy young adult male subjects and multiple oral doses of KM-819 in elderly male subjects.
Time Frame: Part A: Day 1 to 4; Part B: Day 1 to Day 8
Population: All subjects who received at least one dose.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL
  Part A: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
  Part A | 597.5 (140.5) | 1726 (289.7) | 4479 (1423) | 8210 (2912) | 12770 (4321) | 10880 (1108) |  |  |  |  |
  Part B-Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Part B-Day 1 |  |  |  |  |  |  | 1786 (379.4) | 3944 (1453) | 7340 (3890) | 11880 (4525) | 19660 (11160)
  Part B-Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Part B-Day 7 |  |  |  |  |  |  | 1608 (414.2) | 3688 (686.0) | 6333 (2402) | 17330 (10900) | 17020 (5676)

7. Secondary Outcome: AUCinf (Area Under the Plasma Concentration-time Curve From Predose (Time 0) Extrapolated to Infinity)
Description: To evaluate AUCinf of single and multiple ascending oral doses of KM-819 in healthy young adult male subjects and multiple oral doses of KM-819 in elderly male-subjects.
Time Frame: Part A: Day 1 to 4; Part B: Day 1 to Day 8
Population: All subjects who received at least one dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL
  Part A: number analyzed (Participants) | 6 | 6 | 4 | 5 | 5 | 6 | 0 | 0 | 0 | 0 | 0
  Part A | 594.2 (24.4) | 1731 (17.3) | 4872 (30.8) | 7338 (51.9) | 12640 (36.1) | 10970 (9.8) |  |  |  |  |
  Part B-Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0 | 6
  Part B-Day 1 |  |  |  |  |  |  | 1713 (22.4) | 3884 (41.5) | 10070 (30.8) |  | 18550 (57.8)

8. Secondary Outcome: %AUCex (Percentage of AUCinf That is Due to Extrapolation Beyond Tlast)
Description: To evaluate %AUCex of single and multiple ascending oral doses of KM-819 in healthy young adult male subjects and multiple oral doses of KM-819 in elderly male subjects.
Time Frame: Part A: Day 1 to 4; Part B: Day 1 to Day 8
Population: All subjects who received at least one dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
percentage of AUC
  Part A: number analyzed (Participants) | 6 | 6 | 4 | 5 | 5 | 6 | 0 | 0 | 0 | 0 | 0
  Part A | 1.664 (50.5) | 1.331 (51.2) | 1.338 (19.0) | 0.7787 (65.4) | 0.4833 (164.4) | 0.9795 (77.9) |  |  |  |  |
  Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 3 | 0 | 5
  Part B |  |  |  |  |  |  | 1.273 (43.9) | 3.075 (63.3) | 2.263 (84.8) |  | 1.982 (112.1)

9. Secondary Outcome: CL/F (Apparent Oral Clearance)
Description: To evaluate the CL/F of single and multiple ascending oral doses of KM-819 in healthy young adult male subjects and multiple oral doses of KM-819 in elderly male subjects.
Time Frame: Part A: Day 1 to 4; Part B: Day 1 to Day 8
Population: All subjects who received at least one dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
mL/h
  Part A: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
  Part A | 16830 (24.4) | 17340 (17.3) | 20530 (30.8) | 27260 (51.9) | 31650 (36.1) | 18230 (9.8) |  |  |  |  |
  Part B-Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0 | 6
  Part B-Day 1 |  |  |  |  |  |  | 17520 (22.4) | 25740 (41.5) | 19860 (30.8) |  | 10780 (57.8)
  Part B-Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Part B-Day 7 |  |  |  |  |  |  | 19090 (24.8) | 28760 (17.9) | 24930 (7.7) | 20480 (96.4) | 12300 (34.1)

10. Secondary Outcome: Vz/F (Apparent Volume of Distribution)
Description: To evaluate Vz/F of single and multiple ascending oral doses of KM-819 in healthy young adult male subjects multiple oral doses of KM-819 in elderly male subjects.
Time Frame: Part A: Day 1 to 4; Part B: Day 1 to Day 8
Population: All subjects who received at least one dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
mL
  Part A: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
  Part A | 43370 (18.8) | 119800 (23.5) | 271200 (56.6) | 354300 (114.0) | 389300 (49.5) | 277500 (27.3) |  |  |  |  |
  Part B-Day1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0 | 6
  Part B-Day1 |  |  |  |  |  |  | 77710 (32.9) | 201200 (57.6) | 165700 (58.1) |  | 68250 (72.8)
  Part B-Day7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Part B-Day7 |  |  |  |  |  |  | 143400 (33.5) | 241300 (23.6) | 171400 (7.4) | 187100 (151.8) | 88200 (64.9)

11. Secondary Outcome: AUCtau (Area Under the Plasma Concentration-time Curve for a Dosing Interval) (Part B)
Description: To evaluate the pharmacokinetics and pharmacodynamics of single and multiple ascending oral doses of KM-819 in healthy young adult male subjects multiple oral doses of KM-819 in elderly male subjects.
Time Frame: Part B: Day 1 predose (within 30 minutes prior to study drug administration) and 0.25, 0.5, 1, 2, 4, 6, 8, and 12 hours postdose, predose on Days 2, 3, 4, 5, 6, and on Day 7 predose (within 30 minutes prior to study drug administration) and 0.25, 0.5, 1,
Population: All subjects who received at least one dose in Part B
Measure: Mean (Full Range); unit: h*ng/mL
Arm/Group | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*ng/mL | 1612 [1130 to 2320] | 3521 [2760 to 4290] | 8039 [7670 to 8770] | 22830 [11000 to 34700] | 17020 [11000 to 25800]

12. Secondary Outcome: Rac(AUC) (Observed Accumulation by AUC) (Part B)
Description: as for outcome 11
Time Frame: as for outcome 11
Population: All subjects who received at least one dose in Part B
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ratio | 0.8926 [0.70 to 1.13] | 0.9727 [0.69 to 1.37] | 0.7568 [0.57 to 1.00] | 1.485 [0.86 to 2.56] | 0.9241 [0.67 to 1.28]

13. Secondary Outcome: Rac (Cmax) (Observed Accumulation by Cmax) (Part B)
Description: as for outcome 3
Time Frame: as for outcome 11
Population: All subjects who received at least one dose in Part B
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ratio | 0.8173 [0.53 to 1.26] | 1.003 [0.73 to 1.39] | 0.6227 [0.55 to 0.71] | 1.117 [1.00 to 1.25] | 0.9122 [0.53 to 1.58]

14. Secondary Outcome: AUCtau_D (AUCtau Divided by Dose) (Part B)
Description: as for outcome 3
Time Frame: as for outcome 11
Population: All subjects who received at least one dose in Part B
Measure: Mean (Full Range); unit: (h*ng/mL)/mg
Arm/Group | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
(h*ng/mL)/mg | 53.74 [37.7 to 77.4] | 35.21 [27.6 to 42.9] | 40.19 [38.3 to 43.6] | 57.08 [27.5 to 86.6] | 85.09 [55.1 to 129]

15. Secondary Outcome: Change From Baseline for Bond and Lader Visual Analogue Scale (VAS)
Description: The Bond-Lader Visual Analogue Scales (VAS) will be analyzed using 3 factor scores: alertness, contentedness, and calmness. Participants were asked to indicate on the VAS scale ranging from 0 to 100 mm about how they felt at the moment the scale was administered. Baseline is defined as the last available recording prior to dosing on Day 1.
  1. Alertness (Range 0 to 100, the higher scores indicated more alertness)
  2. Mood (Range 0 to 100, where higher scores indicated elevated mood)
  3. Calmness (Range 0 to 100, where higher scores indicated more calmness).
Time Frame: At Day 1 (3 hours post dose), Day2, Day 3, Day 4, and Day 8.
Population: All subjects who received at least one dose.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | Placebo (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B) | Placebo (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 5 | 5 | 6 | 10
units on a scale
  Alertness- Day 1, 3 hours postdose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 5 | 4 | 6 | 10
  Alertness- Day 1, 3 hours postdose | -0.482 (3.6349) | -4.315 (8.8671) | 0.720 (7.2589) | -3.610 (9.4171) | -2.333 (6.4200) | 3.093 (3.7733) | -2.926 (11.4835) | 7.058 (12.2168) | 3.445 (11.1990) | 9.264 (21.4350) | -4.668 (4.6964) | -0.128 (8.7694) | 2.088 (8.4283)
  Alertness-Day 2, 24 hours postdose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 11 | 6 | 6 | 5 | 5 | 6 | 10
  Alertness-Day 2, 24 hours postdose | -3.202 (5.4359) | -0.465 (11.1985) | -2.333 (3.4326) | -0.148 (7.5707) | -2.427 (5.7016) | 2.315 (4.8479) | -0.171 (6.8216) | 0.093 (6.0070) | -5.687 (9.4737) | -0.222 (10.7325) | -0.976 (6.2563) | -3.760 (6.2182) | 0.566 (8.2926)
  Alertness-Day 3, 48 hours postdose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 0 | 0
  Alertness-Day 3, 48 hours postdose | -4.500 (6.2535) | -2.278 (11.9110) | -8.073 (8.6618) | -3.128 (6.5867) | -4.110 (8.6208) | 5.500 (5.2313) | -4.572 (9.7416) |  |  |  |  |  |
  Alertness-Day 4, 72 hours postdose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 0 | 0
  Alertness-Day 4, 72 hours postdose | -6.665 (5.8359) | -3.372 (8.8024) | -6.352 (11.6716) | -6.372 (6.0623) | -3.368 (9.2123) | 3.222 (3.4213) | -7.814 (7.5635) |  |  |  |  |  |
  Calmness-Day 1, 3 hours postdose | 0.42 (8.417) | -3.08 (6.888) | 1.75 (9.832) | -1.17 (9.852) | 0.25 (4.709) | 1.67 (5.279) | -1.04 (6.580) | -10.92 (18.400) | 1.33 (5.654) | -1.00 (36.447) | -12.30 (16.010) | 4.00 (17.593) | 1.40 (6.728)
  Calmness-Day 2, 24 hours postdose | -1.42 (9.952) | 1.00 (9.290) | -3.75 (13.080) | 3.42 (12.064) | 3.92 (3.513) | 0.83 (8.430) | -0.63 (9.033) | -7.33 (18.384) | 0.25 (3.504) | -8.40 (13.093) | -7.70 (20.092) | 8.25 (16.121) | 1.25 (6.233)
  Calmness-Day 3, 48 hours postdose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 0 | 0
  Calmness-Day 3, 48 hours postdose | -5.42 (10.542) | 0.42 (7.651) | -9.92 (9.388) | -2.33 (4.502) | 3.58 (4.188) | 1.00 (5.138) | -3.21 (10.310) |  |  |  |  |  |
  Calmness-Day 4, 72 hours postdose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 0 | 0
  Calmness-Day 4, 72 hours postdose | -3.42 (11.160) | 3.33 (10.567) | -8.50 (11.908) | 1.42 (7.807) | 6.58 (7.249) | 0.42 (4.443) | -2.67 (8.446) |  |  |  |  |  |
  Contentedness-Day 1, 3 hours postdose | -1.83 (6.770) | -2.67 (3.355) | -2.37 (3.194) | -1.33 (1.473) | -1.93 (6.822) | -3.10 (13.121) | 0.90 (6.872) | -1.80 (4.818) | 3.23 (5.251) | 2.52 (18.349) | 0.96 (3.542) | -7.13 (6.565) | -0.42 (3.294)
  Contentedness-Day 2, 24 hours postdose | -7.13 (12.139) | 1.30 (5.383) | -3.53 (3.384) | 1.03 (3.674) | -0.73 (8.911) | -0.53 (9.226) | -1.43 (5.775) | -3.63 (5.126) | -2.23 (5.076) | -5.12 (2.674) | 2.16 (9.459) | -4.43 (5.321) | -1.58 (2.978)
  Contentedness-Day 3, 48 hours postdose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 0 | 0
  Contentedness-Day 3, 48 hours postdose | -7.37 (13.125) | -2.83 (5.159) | -3.80 (5.374) | -1.07 (3.840) | -1.30 (6.549) | 0.37 (7.337) | -2.30 (9.936) |  |  |  |  |  |
  Contentedness-Day 4, 72 hours postdose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 0 | 0
  Contentedness-Day 4, 72 hours postdose | -7.00 (11.021) | -0.80 (2.086) | -3.13 (8.256) | -3.23 (3.024) | -3.93 (5.504) | -1.60 (7.201) | -4.83 (6.200) |  |  |  |  |  |
  Alertness-Day 8, 24 hours postdose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 5 | 5 | 6 | 10
  Alertness-Day 8, 24 hours postdose |  |  |  |  |  |  |  | -2.282 (3.6448) | -8.835 (8.3161) | 3.842 (9.4304) | -7.358 (4.7420) | -6.683 (15.6554) | -2.834 (6.5374)
  Calmness-Day 8, 24 hours postdose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 5 | 5 | 6 | 10
  Calmness-Day 8, 24 hours postdose |  |  |  |  |  |  |  | -7.75 (19.263) | 6.75 (14.754) | 1.90 (7.171) | -6.10 (18.301) | 10.25 (16.825) | 1.40 (10.538)
  Contentedness-Day 8, 24 hours postdose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 5 | 5 | 6 | 10
  Contentedness-Day 8, 24 hours postdose |  |  |  |  |  |  |  | -2.87 (5.731) | -3.27 (2.738) | -0.40 (2.429) | -1.44 (7.249) | -8.27 (8.068) | -1.76 (6.983)

16. Secondary Outcome: Korean Wechsler Adult Intelligence Scale-IV (K-WAIS-IV)
Description: The K-WAIS-IV consists of an assessment of the cognitive ability using a core battery of 10 unique subtests (Block Design, Similarities, Digit Span, Matrix Reasoning, Vocabulary, Arithmetic, Symbol Search, Visual Puzzles, Information, and Coding) that focus on four specific domains of intelligence: verbal comprehension, perceptual reasoning, working memory, and processing speed. The Verbal Comprehension Index, Perceptual Reasoning Index, Working Memory Index, and Processing Speed Index (standard scores: mean=100, standard deviation=15) that are all based on a number of core and supplemental subtests (scaled scores: mean=15, standard deviation=3) that provide pertinent clinical information and flexibility in implementation. The higher values represent a better outcome.
Time Frame: Part A: Day 1; Part B: Day 7
Population: All subjects who received at least one dose
Measure: Mean (Standard Deviation); unit: Intelligence quotient (IQ)
Arm/Group | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | Placebo (Part A) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B) | Placebo (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 10
Intelligence quotient (IQ)
  Day 1, 3 hours postdose | 6.2 (10.05) | -0.3 (8.73) | -3.8 (16.18) | 2.2 (8.04) | 4.8 (6.94) | 3.3 (5.24) | 2.5 (8.87) | 1.7 (5.50) | 4.3 (6.41) | 2.0 (15.12) | 1.2 (4.09) | 1.2 (4.45) | -1.6 (16.19)
  Day 1, 6 hours postdose | 6.5 (14.53) | -1.7 (8.07) | 2.7 (8.43) | 8.7 (9.79) | 6.0 (8.88) | 3.3 (7.50) | 3.3 (7.97) | 3.7 (6.50) | 4.7 (3.72) | 2.2 (7.22) | 0.0 (16.69) | 5.5 (4.97) | 2.9 (13.62)
  Day 1, 12 hours postdose | 12.8 (14.95) | 4.5 (7.82) | 3.0 (14.99) | 10.2 (10.34) | 9.5 (7.66) | 7.3 (5.82) | 4.4 (12.62) | 12.7 (10.39) | 13.2 (4.26) | 11.2 (7.66) | -1.4 (10.21) | 7.0 (5.33) | 6.2 (19.52)
  Day 7, pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 10
  Day 7, pre-dose |  |  |  |  |  |  |  | 10.5 (10.33) | 22.2 (13.29) | 17.6 (6.77) | 11.0 (8.72) | 10.3 (5.57) | 7.3 (19.80)
  Day 7, 3 hours postdose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 10
  Day 7, 3 hours postdose |  |  |  |  |  |  |  | 15.8 (13.88) | 19.7 (6.74) | 24.6 (10.41) | 12.2 (9.76) | 10.2 (5.12) | 6.6 (21.76)
  Day 7, 6 hours postdose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 10
  Day 7, 6 hours postdose |  |  |  |  |  |  |  | 13.7 (21.16) | 27.2 (6.21) | 22.0 (16.32) | 14.8 (12.03) | 12.3 (5.39) | 13.6 (22.47)
  Day 7, 12 hours postdose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 10
  Day 7, 12 hours postdose |  |  |  |  |  |  |  | 17.8 (20.94) | 30.3 (12.48) | 24.4 (9.29) | 18.8 (8.26) | 11.7 (3.78) | 12.8 (20.87)

17. Secondary Outcome: Alpha Synuclein Oligomer in Plasma and CSF (Part B)
Description: To evaluate Alpha synuclein oligomer in plasma and CSF of single and multiple ascending oral doses of KM-819 in healthy young adult male subjects and multiple oral doses of KM-819 in elderly male subjects.
Time Frame: Plasma - Part B: Day 7 (at 1 hour after last dosing) / CSF - Part B: Day 7 (at 1 hour after last dosing)
Population: All subjects who received at least one dose in Part B
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B) | Placebo (Part B)
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 6 | 10
pg/mL
  CSF, Day 7, 1 hour postdose | 49.9424 [1.118 to 188.833] | -252.5578 [-1565.068 to 47.610] | 0.6012 [-25.141 to 24.998] | 18.2112 [-121.943 to 163.679] | 34.8672 [-22.683 to 95.017] | 20.3025 [-82.488 to 145.654]
  Plasma, Day 7, 1 hour postdose | 3884.4127 [-40474.448 to 47672.249] | 575.4570 [-29995.002 to 27948.723] | 3809.5090 [-16201.393 to 18993.995] | -64843.287 [-297443.64 to 4664.264] | -11712.090 [-45482.537 to 880.845] | -4464.9082 [-24410.549 to 23915.230]

18. Secondary Outcome: Change From Baseline Total Tau in CSF (Part B)
Description: To evaluate Total Tau in CSF of single and multiple ascending oral doses of KM-819 in healthy young adult male subjects and multiple oral doses of KM-819 in elderly male subjects.
Time Frame: CSF - Part B: Day 1 (at -120 minutes to 0 minute prior to the first dosing) and on Day 7 (at 1 hour after last dosing)
Population: All subjects who received at least one dose in Part B
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B) | Placebo (Part B)
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 6 | 10
pg/mL | 60.3043 [-23.213 to 145.209] | 9.2313 [-9.048 to 33.901] | -3.1593 [-15.058 to 22.546] | 27.8648 [-32.813 to 134.771] | 29.2961 [-52.079 to 203.508] | 20.8198 [-13.358 to 82.099]

19. Secondary Outcome: Change From Baseline Phospho-Tau in CSF (Part B)
Description: To evaluate Phospho-Tau of single and multiple ascending oral doses of KM-819 in healthy young adult male subjects and multiple oral doses of KM-819 in elderly male subjects.
Time Frame: CSF - Part B: Day 1 (at -120 minutes to 0 minute prior to the first dosing) and on Day 7 (at 1 hour after last dosing)
Population: All subjects who received at least one dose in Part B
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B) | Placebo (Part B)
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 6 | 10
pg/mL | 6.4132 [-13.590 to 42.811] | 0.2072 [-1.154 to 2.231] | 4.4672 [-1.534 to 18.292] | 6.7032 [-2.773 to 19.666] | 5.1606 [-5.717 to 23.325] | 5.3123 [-3.592 to 23.931]

20. Secondary Outcome: Ratio of CSF Concentration/Plasma Cmax (Part B)
Description: Ratio of CSF concentration/Plasma Cmax
Time Frame: Plasma - Part B: Day 7 (at 1 hour after last dosing) / CSF - Part B: on Day 7 (at 1 hour after last dosing)
Population: All subjects who received at least one dose in Part B
Measure: Mean (Full Range); unit: Ratio
Arm/Group | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
Number analyzed (Participants) | 3 | 3 | 4 | 5
Ratio | 0.00067004 [0.00040485 to 0.00085699] | 0.00074179 [0.00047881 to 0.00090404] | 0.00048832 [0.00011022 to 0.0013316] | 0.00031749 [0.00018612 to 0.00045000]

ADVERSE EVENTS:
Time Frame: From screening (Day-28 to Day -2), Day -1 to Day 4, Day 7, and follow-up visit Day 14.
Description: An AE is any untoward medical occurrence that occurs in a subject or clinical investigation subject administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment.
Arm/Group | Placebo (Part A) | KM-819 - 10 mg (Part A) | KM-819 - 30 mg (Part A) | KM-819 - 100mg (Part A) | KM-819 200mg (Part A) | KM-819 - 400mg (Part A) | KM-819 200mg (Elderly Male Subjects) (Part A) | Placebo (Part B) | KM-819 30 mg (Part B) | KM-819 100 mg (Part B) | KM-819 200mg (Part B) | KM-819 400mg (Part B) | KM-819 200mg (Elderly Male Subjects) (Part B)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/6 | 0/6 | 1/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/12 | 2/6 | 2/6 | 3/6 | 1/6 | 0/6 | 4/6 | 10/10 | 6/6 | 5/6 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part A) (N=12) | KM-819 - 10 mg (Part A) (N=6) | KM-819 - 30 mg (Part A) (N=6) | KM-819 - 100mg (Part A) (N=6) | KM-819 200mg (Part A) (N=6) | KM-819 - 400mg (Part A) (N=6) | KM-819 200mg (Elderly Male Subjects) (Part A) (N=6) | Placebo (Part B) (N=10) | KM-819 30 mg (Part B) (N=6) | KM-819 100 mg (Part B) (N=6) | KM-819 200mg (Part B) (N=6) | KM-819 400mg (Part B) (N=6) | KM-819 200mg (Elderly Male Subjects) (Part B) (N=6)
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — 1 patient had a headache which was considered unlikely to be related to KM-819, and probably related to the lumbar puncture procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=12) | KM-819 - 10 mg (Part A) (N=6) | KM-819 - 30 mg (Part A) (N=6) | KM-819 - 100mg (Part A) (N=6) | KM-819 200mg (Part A) (N=6) | KM-819 - 400mg (Part A) (N=6) | KM-819 200mg (Elderly Male Subjects) (Part A) (N=6) | Placebo (Part B) (N=10) | KM-819 30 mg (Part B) (N=6) | KM-819 100 mg (Part B) (N=6) | KM-819 200mg (Part B) (N=6) | KM-819 400mg (Part B) (N=6) | KM-819 200mg (Elderly Male Subjects) (Part B) (N=6)
Eye swelling (Eye disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 (2) | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0
Influenza (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 2 (2) | 2 (4) | 2 (3) | 1 (2) | 5 (11) | 4 (7) | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 2 (2) | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 1 (1) | 4 (5) | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 4 (4) | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 (3) | 0 | 2 (2) | 1 (1) | 1 (2) | 2 (3)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (2) | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT03022799/Prot_000.pdf
  • Informed Consent Form (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT03022799/ICF_001.pdf
  • Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT03022799/SAP_002.pdf